CLINICAL TRIAL: NCT02855918
Title: Modification of the Expression of ADARs and PDE8A Editing in Suicidal Behavior
Brief Title: Blood Biomarkers in Suicidal Behaviour
Acronym: 2BSB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Sys2Diag, Mixt laboratory CNRS/Alcediag, Montpellier (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UF 9625; 2015-A01978-41 (Other: Agence Nationale de Sécurité des Médicaments)
Record Dates: First submitted 2016-07-15; First posted 2016-08-04 (Estimated); Last update posted 2021-12-27 (Actual); Status verified 2021-12

CONDITIONS: Major Depression
Keywords: Psychiatry; Depressive disorder; Suicidal behavior; Genetics
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Blood sample for genetic purpose (Other): All the participants performed the same evaluations and blood analysis.
  The study is composed of 3 groups :
  * depressed patients with an history of suicide attempt
  * depressed patients without any history of suicide attempt
  * healthy controls without any history of psychopathology
  Interventions: Other: Blood sample for genetic purpose

INTERVENTIONS:
Other: Blood sample for genetic purpose — All the participants will performed the same evaluations and blood analysis :
  * A clinical assessment by psychiatrist
  * Self report questionnaires for the assessment of a potential mood disorder and history of SB, moral/physical pain, personality traits…
  * A neuropsychological assessment for the evaluations of cognitive performances
  * A routine blood sampling to the realization of a standard blood test
  * A specific blood sampling (PAXgene® tubes) to extract total RNA of blood cells and measure the expression of ADARS RNA and editing of the PDE8A transcript.

SUMMARY:
Suicidal behavior (SB) is a major public health problem in France, with more than 10,000 suicides and 220,000 suicide attempts per year.

According to the commonly accepted model for understanding suicidal behavior, individuals who carry a suicidal act when subjected to stress factors (environmental stress, depression, substance ...) are those which have a specific vulnerability.

These vulnerabilities can be considered as clinical parameters (propensity to despair, aggressive and/or impulsive traits), neurobiological parameters (dysfunction of the serotonergic system, ...) and cognitive parameters (taking disadvantageous decision ...). Suicidal vulnerability is partly underpinned by genetic factors. The interest of current researches is to identify biomarkers that will improve the opportunities for early identification of subject with a risk for SB. Numerous scientific studies, including post-mortem studies of the brains of suicide completers, have established a link between dysregulation of the ribonucleic acids editing (RNA) of certain genes, the enzymatic activity of Adenosine deaminases acting on RNA (ADARS) responsible for this edition and suicidal behavior. A prospective study is needed to quantify and qualify in the blood of depressed patients (with or without a history of suicide) and healthy controls, the editing changes and the expression and alteration of the activity of ADARS.

DETAILED DESCRIPTION:
Over two years, 600 participants will be recruited:

* 225 subjects with current major depressive episode and an history of suicide attempt (depressed suicide attempters)
* 225 subjects with current major depressive episode but with no personal history of suicide attempt (affective controls)
* 150 subjects with no history of psychopathology whole life (healthy controls)

Each patient will attend a total of 3visits during a follow-up period of 6 months +/- 15 days (inclusion, visit at 3 and 6 months).

ELIGIBILITY:
No specific inclusion criteria :

* 18 to 65 years
* Subject who signed the informed consent
* Able to understand the nature, purpose and methodology of the study
* Able to understand and perform the clinical and neuropsychological evaluations.

Specific inclusion criteria depressed suicide attempters:

* Subject whose primary psychiatric diagnosis is a major depressive episode according to Diagnostic and Statistical Manual of Mental Disorders -5 (DSM-5) criteria
* Personal history of suicide attempt

affective controls:

* Subject whose primary psychiatric diagnosis is a major depressive episode according to DSM-5 criteria
* No personal history of suicide attempt

healthy controls:

* No personal history of psychiatric disorders (Axis I ) defined by the Mini International Neuropsychiatric Interview (MINI) according to the DSM-5 criteria
* No history of suicide attempt

Exclusion criteria

* Refusal of participation
* Deprived of liberty Subject (by judicial or administrative decision)
* Subject protected by law (guardianship)
* Subject exclusion period in relation to another protocol
* Subject is not affiliated to a social security scheme, beneficiary or not such a plan
* Subject for which the maximum annual amount of allowances of € 4,500 has been reached
* Pregnant women
* Breastfeeding Women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2016-09-23 (Actual); Primary Completion 2020-06-24 (Actual); Study Completion 2020-06-24 (Actual)

PRIMARY OUTCOMES:
Evolution of the modification of the expression of Adenosine deaminases acting on RNA (ADARs) and of the editing profile of phospho-diesterase 8A (PDE8A) | At the inclusion visit, 3 months and 6 months after the inclusion
  Studying ADARs expression and RNA editing of genes associated with SB, including PDE8A and comparison of these results between healthy controls and depressed patients with or without history of SB

SECONDARY OUTCOMES:
Modification of the expression of ADAR1a enzymes | At the inclusion visit, 3 months and 6 months after the inclusion
  Comparison of the profiles of ADARs expression and PDE8A editing between non suicidal and suicidal depressed patients and healthy controls
Modification of the expression and RNA editing of Spindle And Kinetochore Associated protein 2 (SKA2) | At the inclusion visit, 3 months and 6 months after the inclusion
  Comparison between non suicidal and suicidal depressed patients and healthy controls
Modification of the expression of ADAR1b enzymes | At the inclusion visit, 3 months and 6 months after the inclusion
  Comparison of the profiles of ADARs expression and PDE8A editing between non suicidal and suicidal depressed patients and healthy controls
Modification of the expression of ADAR2 enzymes | At the inclusion visit, 3 months and 6 months after the inclusion
  Comparison of the profiles of ADARs expression and PDE8A editing between non suicidal and suicidal depressed patients and healthy controls
Modification of the expression and RNA editing of Spermidine/Spermine N1-Acetyltransferase 1 (SAT1) | At the inclusion visit, 3 months and 6 months after the inclusion
  Comparison between non suicidal and suicidal depressed patients and healthy controls
Modification of the expression and RNA editing of Interleukins (ILs) | At the inclusion visit, 3 months and 6 months after the inclusion
  Comparison between non suicidal and suicidal depressed patients and healthy controls
Modification of the expression and RNA editing of Chemokines (CXCLs) | At the inclusion visit, 3 months and 6 months after the inclusion
  Comparison between non suicidal and suicidal depressed patients and healthy controls
Modification of the expression and RNA editing of Brain derived Neurotrphic factor (BDNF) | At the inclusion visit, 3 months and 6 months after the inclusion
  Comparison between non suicidal and suicidal depressed patients and healthy controls
Modification of the expression and RNA editing of Cluster of differentiation 24 (CD24) | At the inclusion visit, 3 months and 6 months after the inclusion
  Comparison between non suicidal and suicidal depressed patients and healthy controls
Modification of the expression and RNA editing of Three prime repair exonuclease 1 (TREX1) | At the inclusion visit, 3 months and 6 months after the inclusion
  Comparison between non suicidal and suicidal depressed patients and healthy controls
Modification of the expression and RNA editing of Interferon stimulated gene 15 (ISG15) | At the inclusion visit, 3 months and 6 months after the inclusion
  Comparison between non suicidal and suicidal depressed patients and healthy controls
Modification of the expression and RNA editing of Tumor necrosis factor alpha (TNF alpha) | At the inclusion visit, 3 months and 6 months after the inclusion
  Comparison between non suicidal and suicidal depressed patients and healthy controls
Modification of the expression and RNA editing of Vascular endothelial growth factor (VEGF) | At the inclusion visit, 3 months and 6 months after the inclusion
  Comparison between non suicidal and suicidal depressed patients and healthy controls
Modification of the expression and RNA editing of Hydroxytryptamine receptor 2A (HTR2A) | At the inclusion visit, 3 months and 6 months after the inclusion
  Comparison between non suicidal and suicidal depressed patients and healthy controls
Modification of the expression and RNA editing of insulin-like growth factor protein 7 (IGFB7) | At the inclusion visit, 3 months and 6 months after the inclusion
  Comparison between non suicidal and suicidal depressed patients and healthy controls

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Montpêllier, France

IPD SHARING:
Plan to Share IPD: No